CLINICAL TRIAL: NCT02177266
Title: Colchicine Versus Placebo in Post-Cardiac Surgery Patients to Prevent Post-Pericardiotomy Syndrome and Atrial Fibrillation
Brief Title: Colchicine to Prevent Post-Pericardiotomy Syndrome and Atrial Fibrillation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in recruiting patients
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jae K. Oh, M.D., Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-008553
Record Dates: First submitted 2014-06-18; First posted 2014-06-27 (Estimated); Results first posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-05

CONDITIONS: Atrial Fibrillation; Post-pericardiotomy Syndrome; Constriction
MeSH Terms: conditions — Atrial Fibrillation; Postpericardiotomy Syndrome; Constriction, Pathologic | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): A placebo pill (identical to the study drug Colchicine) will be given in a double-blinded fashion to study participants randomized to placebo.
  Interventions: Drug: Placebo
- Colchicine (Experimental): Colchicine 0.6mg bid will be given to study participants randomized to the study drug arm beginning at 48-72 hours prior to the planned cardiac surgery and then continued for a total of 30 days.
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — Colchicine 0.6mg bid will be given to study participants randomized to the study drug arm beginning at 48-72 hours prior to the planned cardiac surgery and then continued for a total of 30 days.
  Other Names: Colcrys
  Arms: Colchicine
Drug: Placebo — The placebo will match the study drug.
  Arms: Placebo

SUMMARY:
The study will determine the benefit of Colchicine versus placebo for cardiac surgery patients on the post-operative development of atrial fibrillation and post-pericardiotomy syndrome.

Primary Objective. Colchicine will reduce the composite endpoint of incidence of post-operative atrial fibrillation and post-pericardiotomy syndrome at 3 months following cardiac surgery.

Secondary Objectives.

1. Colchicine will reduce the incidence of constrictive physiology on echocardiography at 3 months following cardiac surgery.
2. Reduction in the burden of symptomatic and asymptomatic atrial fibrillation in the 3 months following cardiac surgery with the use of colchicine.

DETAILED DESCRIPTION:
Background. Patients undergoing cardiac surgery are at risk for post-pericardiotomy syndrome and post-operative atrial fibrillation. It is unknown whether post-pericardiotomy syndrome predisposes patients to constrictive pericarditis, but cardiac surgery is currently the most common cause of constrictive pericarditis. A multicenter European study demonstrated that Colchicine is a promising treatment to help prevent the development of pericardial effusions, atrial fibrillation and post-pericardiotomy syndrome. However, Colchicine is not routinely given to patients after a cardiac surgery and the impact of Colchicine on post-operative atrial fibrillation and constrictive pericarditis have not been studied in the United States.

Methods. This is a randomized, double-blinded placebo controlled study for patients undergoing cardiac surgery to determine if Colchicine in comparison to placebo is effective in preventing the development of post-operative atrial fibrillation, post-pericardiotomy syndrome and constrictive physiology. The investigators will randomize 278 adults prior to undergoing cardiac surgery for coronary artery bypass graft (CABG) or aortic valve disease to receive either placebo or Colchicine 0.6mg bid for one month starting 48-72 hours preoperatively. The investigators will follow participants for 3 months to determine the development of a post-pericardiotomy syndrome. In addition, post-operative atrial fibrillation will be determined based on continuous telemetry from operation up to 5 days prior to hospital discharge and after discharge by using remote telemetry monitoring with BodyGuardianTM. C-reactive protein (CRP) will be obtained prior to hospital discharge and at 3 month follow-up. Echocardiography will be done initially in the post-operative course prior to hospital discharge and then again at 3 months to assess for the presence of pericardial effusion, diastolic dysfunction, left atrial enlargement and constrictive physiology. The presence of pleural effusion will be done by echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult patients (age > 40) undergoing standard (non-minimally invasive) coronary artery bypass surgery and/or aortic valve surgery will be approached for enrollment.
* All patients must be able to provide informed consent and comply with the 3 month follow-up.
* For women of reproductive capability, contraception is necessary and required.

Exclusion Criteria:

* Epidermal growth factor receptor (eGFR) < 30 mL/min/1.73 m^2, serum creatinine > 2.5 mg/dL or requiring dialysis
* Known permanent or current atrial fibrillation (history of paroxysmal atrial fibrillation allowed if in sinus rhythm at present)
* Allergy to colchicine or already treated with colchicine.
* Known blood dyscrasia (acute or chronic leukemia, pancytopenia, aplastic anemia, leukopenia)
* Known serious gastrointestinal disease
* Known severe liver disease (cirrhosis, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2x the upper limit of normal, Model End Stage Liver Disease (MELD) score > 20)
* Women of childbearing potential not using contraception.
* Patients with HIV or AIDS as the use of protease inhibitors can result in serious colchicine toxicity.
* Patients who are treated with strong CYP3A4 inhibitors (clarithromycin/erythromycin, chloramphenicol, ketoconazole/itraconazole, and nefazodone).
* There is a risk of rhabdomyolysis with the use of digoxin and colchicine, we will exclude patients who require ongoing treatment with digoxin.
* Inability or unwillingness of the individual to give written informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Oh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Placebo | Colchicine
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Colchicine | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Post Cardiac Surgery Atrial Fibrillation or Post-pericardiotomy Syndrome.
Time Frame: Baseline to 3 months
Population: The data were not analyzed because the 2 subjects enrolled withdrew before completing the study; the study was terminated early due to the difficulty in enrolling subjects.
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Trans-thoracic Echocardiography for Constriction
Time Frame: Baseline to 3 months
Population: as for outcome 1
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Time Frame: Baseline - 3 months
Population: as for outcome 1
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Placebo | Colchicine
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1) | Colchicine (N=1)
Skin breakdown (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Reaction to remote telemetry monitoring device (BodyGuardian).
Nausea and dry heaves (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The data were not analyzed because the 2 subjects enrolled withdrew before completing the study; the study was terminated early due to the difficulty in enrolling subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes